CLINICAL TRIAL: NCT03433703
Title: A Single-Arm, Multicenter, Phase 2 Trial to Evaluate Safety and Efficacy of Treatment of Physician Choice (TPC) Following First-Line Treatment of Lenvatinib in Subjects With Unresectable Hepatocellular Carcinoma (uHCC)
Brief Title: Trial to Evaluate Safety and Efficacy of Treatment of Physician Choice (TPC) Following First-Line Treatment of Lenvatinib in Subjects With Unresectable Hepatocellular Carcinoma (uHCC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study recruitment was stopped due to difficulty in enrolling the targeted number of participants.
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7080-M001-222
Record Dates: First submitted 2018-02-09; First posted 2018-02-14 (Actual); Results first posted 2019-12-06 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2018-06

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Unresectable hepatocellular carcinoma; Lenvatinib; E7080
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lenvatinib (Experimental): Participants will receive lenvatinib 12 or 8 milligrams (mg) once daily in continuous 28-day cycles until disease progression, development of unacceptable toxicity, participant request, withdrawal of consent, or study termination by the sponsor. Upon completion of lenvatinib treatment, eligible participants will receive commercially available systemic TPC for hepatocellular carcinoma in the subsequent treatment period.
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib capsules will be administered orally, once daily in continuous 28-day cycles.
  Body weight (BW) ≥60 kilograms (kg) - Lenvatinib 12 mg (taken as three 4-mg capsules); BW <60 kg - Lenvatinib 8 mg (taken as two 4-mg capsules)
  Other Names: LENVIMA®; E7080

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of subsequent systemic treatment of physician's choice (TPC) following the first-line lenvatinib treatment in unresectable hepatocellular carcinoma (uHCC) participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants must have confirmed diagnosis of unresectable Hepatocellular Carcinoma (uHCC) with any of the following criteria:

  1. Histologically or cytologically confirmed diagnosis of uHCC
  2. Clinically confirmed diagnosis of uHCC according to American Association for the Study of Liver Diseases criteria, including cirrhosis of any etiology or with chronic hepatitis B or C infection criteria
* At least one measurable target lesion regardless if hepatic or non-hepatic according to modified Response Evaluation Criteria in Solid Tumors (mRECIST) meeting the following criteria:

  1. Hepatic lesion

     * The lesion can be accurately measured in at least one dimension as ≥1.0 centimeters (cm) (viable tumor for typical; and longest diameter for atypical), and
     * The lesion is suitable for repeat measurement,
  2. Nonhepatic lesion

     * Lymph node lesion that measures at least one dimension as ≥1.5 cm in the short axis
     * Non-nodal lesion that measures ≥1.0 cm in the longest diameter Lesions previously treated with radiotherapy or locoregional therapy must show radiographic evidence of disease progression to be deemed a target lesion.
* Participants categorized on the Barcelona Clinic Liver Cancer staging system to Stage B (not applicable for transarterial chemoembolization) or Stage C
* Adequate bone marrow function, liver function, blood coagulation function, renal function, and pancreatic function as assessed by laboratory tests.
* Adequately controlled blood pressure (BP) with up to 3 antihypertensive agents, defined as BP ≤150/90 millimeters of mercury (mmHg) at Screening and no change in antihypertensive therapy within 1 week prior to Cycle 1/Day 1
* Child-Pugh A
* Eastern Cooperative Oncology Group Performance Status of 0 or 1
* Survival expectation of 12 weeks or longer before starting study drug

Key Exclusion Criteria:

* Imaging findings for HCC corresponding to any of the following:

  1. HCC with ≥50% liver occupation
  2. Clear invasion into the bile duct
  3. Portal vein invasion at the main portal branch (Vp4)
* Participants who have received any systemic chemotherapy, including sorafenib, regorafenib or other anti-vascular endothelial growth factor therapy, nivolumab, or any systemic investigational anticancer agents, including lenvatinib, for advanced/uHCC.
* Participants who have received any anticancer therapy (including surgery, percutaneous ethanol injection, radio frequency ablation, transarterial [chemo] embolization, hepatic intra-arterial chemotherapy, biological, immunotherapy, hormonal, or radiotherapy) or any blood enhancing treatment (including blood transfusion, blood products, or agents that stimulate blood cell production, e.g., granulocyte colony-stimulating factor) within 28 days prior to the first dose of lenvatinib study treatment.
* Participants who have not recovered from toxicities as a result of prior anticancer therapy such as the local hepatic injection chemotherapy or any prior therapy for other cancer types.
* Significant cardiovascular impairment within 6 months of the first dose of study drug
* Prolongation of QT interval corrected for heart rate using Fridericia's correction (QTcF) to >480 milliseconds (ms)
* Gastrointestinal malabsorption or any other condition that might affect the absorption of lenvatinib in the opinion of the investigator
* Bleeding or thrombotic disorders or use of anticoagulants such as warfarin or similar agents requiring therapeutic international normalized ratio monitoring
* Gastrointestinal bleeding event or active hemoptysis (bright red blood of at least half teaspoon) within 28 days prior to the first dose of lenvatinib study treatment
* Gastric or esophageal varices that require treatment
* Active malignancy (except for HCC or definitively treated melanoma in-situ, basal or squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix) within the past 36 months
* Any history of or current brain or subdural metastases
* Participants having >1+ proteinuria on urine dipstick testing will undergo 24-hour urine collection for quantitative assessment of proteinuria. Participants with urine protein ≥1 grams/24 hour will be ineligible
* Arterial-portal venous shunt or arterial-venous shunt preventing proper diagnosis of tumor
* Any medical or other condition that in the opinion of the investigator would preclude the participant's participation in a clinical study
* Known intolerance to lenvatinib or any of the excipients
* Human immunodeficiency virus positive or active infection requiring treatment (except for hepatitis virus)
* Any history of drug or alcohol dependency or abuse within the prior 2 years
* Major surgery within 3 weeks prior to the first dose of lenvatinib study treatment or scheduled for surgery during the study
* Participant has had a liver transplant
* Females who are breastfeeding or pregnant at Screening or Baseline
* Females of childbearing potential who within 28 days before study entry did not use a highly effective method of contraception or do not agree to use a highly effective method of contraception throughout the entire study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2019-01-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - California Liver Research Institute, Pasadena, California
  - University of Florida, Gainesville, Florida
  - University of Louisville, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 3 investigative sites in the United States from 26 April 2018 to 07 January 2019.
Pre-assignment Details: A total of 8 participants were enrolled, of these, 6 were screen failures and 2 were treated. Upon completion of lenvatinib treatment, eligible participants were to receive commercially available systemic treatment of physician choice (TPC). However, because of early termination of study no participants received TPC.
Groups:
- Lenvatinib: Participants received lenvatinib 8 or 12 milligram (mg), capsule, orally, once daily in 28 day continuous cycles until disease progression (PD), development of unacceptable toxicity, participant request, withdrawal of consent, or study termination by the sponsor. Body weight (BW) greater than or equal to (>=) 60 kilograms (kg) - lenvatinib 12 mg (taken as three 4 mg capsules); BW less than (<) 60 kg - lenvatinib 8 mg (taken as two 4 mg capsules).
Period: Overall Study
Arm/Group | Lenvatinib
Started | 2
Completed | 0
Not Completed | 2
Not completed — Study terminated by Sponsor | 2

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set (Full Analysis Set) included all participants who received at least 1 dose of the lenvatinib treatment.
Groups:
- Lenvatinib: Participants received lenvatinib 8 or 12 mg, capsule, orally, once daily in 28 day continuous cycles until PD, development of unacceptable toxicity, participant request, withdrawal of consent, or study termination by the sponsor. BW >=60 kg - lenvatinib 12 mg (taken as three 4 mg capsules); BW <60 kg - lenvatinib 8 mg (taken as two 4 mg capsules).
Arm/Group | Lenvatinib
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: From the first dose of study drug up to 28 days after the last dose of study drug (approximately 3 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib
Number analyzed (Participants) | 2
Participants
  TEAEs | 1
  SAEs | 1

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of first dose of study treatment to the date of death from any cause. Participants who are lost to follow-up are censored at the last date the participant was known to be alive, and participants who remain alive are censored at the time of data cutoff. OS was to be calculated using Kaplan-Meier estimate and presented with 2-sided 95% confidence interval.
Time Frame: From first dose date until date of death from any cause (approximately 3 months)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib
Number analyzed (Participants) | 2
months | NA [NA to NA] — Data from pre-specified Kaplan Meier estimation cannot be reported, because of insufficient number of participants with events.

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS based on modified Response Evaluation Criteria in Solid Tumors (mRECIST) (and including the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 conventions for non-hepatic lesions) is defined as the time from the date of the first dose of first-line lenvatinib treatment to the date of the first documentation of PD, or the date of death during the subsequent systemic TPC, whichever occurs first. PD is defined at least 20% increase (including an absolute increase of at least 5 millimeter [mm]) in the sum of diameters of target lesions, taking as reference the smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions. PFS was to be calculated using Kaplan-Meier estimate and presented with 2-sided 95% confidence interval.
Time Frame: From first dose date until PD or date of death from any cause (approximately 3 months)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib
Number analyzed (Participants) | 2
months | NA [NA to NA] — Data from pre-specified Kaplan Meier estimation cannot be reported, because of insufficient number of participants with events.

4. Secondary Outcome: Time to Progression (TTP)
Description: TTP based on mRECIST (and including the RECIST 1.1 conventions for non-hepatic lesions) is defined as the time from the date of the first dose of first-line lenvatinib treatment to the date of the first documentation of disease progression during subsequent systemic TPC. PD is defined at least 20% increase (including an absolute increase of at least 5 mm) in the sum of diameters of target lesions, taking as reference the smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions. TTP was to be calculated using Kaplan-Meier estimate and presented with 2-sided 95% confidence interval.
Time Frame: From first dose date until PD (approximately 3 months)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib
Number analyzed (Participants) | 2
months | NA [NA to NA] — Data from pre-specified Kaplan Meier estimation cannot be reported, because of insufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 28 days after the last dose of study drug (approximately 3 months)
Arm/Group | Lenvatinib
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenvatinib (N=2)
Hepatic encephalopathy (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenvatinib (N=2)
Urinary tract infection (Infections and infestations) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
The study was terminated due to difficulty in enrolling the targeted number of participants. Secondary endpoints could not be analyzed because of very low sample size. No safety concerns involved in decision to stop enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-24): https://cdn.clinicaltrials.gov/large-docs/03/NCT03433703/Prot_SAP_000.pdf